CLINICAL TRIAL: NCT00268320
Title: Clinical Investigation of the Medtronic Concerto™ Cardiac Resynchronization Therapy (CRT) and Implantable Cardioverter Defibrillator (ICD) Therapies (CRT+ICD Device)
Brief Title: Clinical Investigation of the Medtronic Concerto™ Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 230
Record Dates: First submitted 2005-12-21; First posted 2005-12-22 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Congestive Heart Failure, Atrial Arrhythmia, Atrial Tachyarrhythmia, Atrial Fibrillation
Keywords: congestive heart failure, atrial arrhythmia, cardiac resynchronization therapy, implantable cardioverter defibrillator
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy+Implantable Cardioverter Defibrillator

SUMMARY:
Heart failure is a progressive disease that decreases the pumping action of the heart. This may cause a backup of fluid in the heart and may result in heart beat changes. When there are changes in the heart beat sometimes an implantable heart device is used to control the rate and rhythm of the heart beat. In certain heart failure cases, when the two lower chambers of the heart no longer beat in a coordinated manner, cardiac resynchronization therapy may be prescribed.

People who have a dangerously fast heart beat, or whose heart is at risk of stopping beating, may be in need of an electronic device called an implantable cardioverter defibrillator (ICD).

Atrial tachyarrhythmia (AT) is the name for rapid beats in the upper chambers of the heart. People with AT may experience symptoms such as heart palpitations (a racing or pounding feeling in the chest), shortness of breath, dizziness, fatigue or weakness.

The purpose of this study is to study an investigational implantable device containing Cardiac Resynchronization Therapy (CRT) and Implantable Cardioverter Defibrillator (ICD) therapies (CRT+ICD device) in subjects who are at significant risk of developing atrial tachyarrhythmias.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who require the implantation of an Implantable Cardioverter Defibrillator
* Subjects who have heart failure that severely limits daily activities (NYHA Class III) or Subjects who have severe heart failure and should always be resting (NYHA Class IV)
* Subjects with reduced heart pumping function (left ventricular ejection fraction ≤ 35%)

Exclusion Criteria:

* Subjects who have constant atrial fibrillation (top chambers of the heart beat too fast continuously)
* Subjects who are post-heart transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270
Dates: Start 2006-01; Primary Completion 2006-06 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Complication rate
Atrial defibrillation effectiveness

SECONDARY OUTCOMES:
Change in patient health status during the study
System performance
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Not required for IDE studies
Locations (51):
- United States (30):
  - Anchorage, Alaska
  - Phoenix, Arizona
  - Santa Monica, California
  - Jacksonville, Florida
  - Orlando, Florida
  - Pensacola, Florida
  - Atlanta, Georgia
  - Evanston, Illinois
  - Fort Wayne, Indiana
  - Des Moines, Iowa
  - Brighton, Massachusetts
  - Detroit, Michigan
  - Saint Paul, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Newark, New Jersey
  - Albuquerque, New Mexico
  - Syracuse, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Pittsburgh, Pennsylvania
  - West Reading, Pennsylvania
  - Charleston, South Carolina
  - Nashville, Tennessee
  - Austin, Texas
  - Fort Worth, Texas
  - Richmond, Virginia
  - Tacoma, Washington
  - Morgantown, West Virginia
- Austria (2):
  - Linz
  - Sankt Pölten
- Copenhagen, Denmark
- Germany (6):
  - Aachen
  - Bernau
  - Bochum
  - Göttingen
  - Heidelberg
  - Münster
- Pátrai, Greece
- Italy (2):
  - Negrar, Veneto
  - Bologna
- Japan (3):
  - Tsukuba, Ibaraki
  - Suita, Osaka
  - Shinjuku-ku, Tokyo
- Netherlands (2):
  - Eindhoven
  - Rotterdam
- Oslo, Norway
- Valencia, Spain
- Basel, Switzerland
- Southhampton, United Kingdom